CLINICAL TRIAL: NCT03553407
Title: Evaluation of the Analgesic Effect of Low Intensity Laser in Patients With Pulpitis of Mandibular Molars. Randomized, Double Blind Study.
Brief Title: Analgesic Effect of Low Intensity Laser in Patients With Pulpitis of Mandibular Molars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Isabel Peixoto Tortamano, professor of the department of stomatology of the university of sao paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser
Record Dates: First submitted 2017-12-12; First posted 2018-06-12 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pulpitis - Irreversible
Keywords: Low level laser; Pulpitis; Mandibular molars
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Level Laser - Pulse (Experimental): In this group the patient will receive the following laser protocol: 880nm, 30mW, 3.6 J / cm², 25 Hz
  Interventions: Device: Low Level Laser - Pulse
- Low Level Laser - continuous (Experimental): In this group the patient will receive the following laser protocol: 880nm, 30mW, 3.6 J / cm²
  Interventions: Device: Low Level Laser - continuous
- Low Level Laser - Placebo (Placebo Comparator): In this group the patient will receive the protocol with the equipment turned off.
  Interventions: Device: Low Level Laser - placebo

INTERVENTIONS:
Device: Low Level Laser - Pulse — The laser will be applied at a single point in contact, perpendicular to the surface of the tooth in a region that presents healthy enamel, towards the pulp chamber. The laser chosen was the low power diode laser with the following protocols: Group 1 (880nm, 30mW, 3.6 J / cm², 25 Hz) and Group 2 (880nm, 30mW, 3.6 J / cm²), after 10 minutes we will ask to the patient again from 0 to 3 the level of pain, to then proceed to the anesthetic phase.
  Arms: Low Level Laser - Pulse
Device: Low Level Laser - continuous — The laser will be applied at a single point in contact, perpendicular to the surface of the tooth in a region that presents healthy enamel, towards the pulp chamber. The laser chosen was the low power diode laser with the following protocols: Group 1 (880nm, 30mW, 3.6 J / cm², 25 Hz) and Group 2 (880nm, 30mW, 3.6 J / cm²), after 10 minutes we will ask to the patient again from 0 to 3 the level of pain, to then proceed to the anesthetic phase.
  Arms: Low Level Laser - continuous
Device: Low Level Laser - placebo — placebo will be applied at a single point in contact, perpendicular to the surface of the tooth in a region that presents healthy enamel, towards the pulp chamber. The laser chosen was the low power diode laser with the following protocols: Group 1 (880nm, 30mW, 3.6 J / cm², 25 Hz) and Group 2 (880nm, 30mW, 3.6 J / cm²), after 10 minutes we will ask to the patient again from 0 to 3 the level of pain, to then proceed to the anesthetic phase.
  Arms: Low Level Laser - Placebo

SUMMARY:
The present study has the objective of evaluating whether the previous therapy with low intensity laser, through its analgesic effect, can promote a greater comfort specifically for patient with pulpitis in mandibular molars. 75 patients with pain from mandibular molar pulpitis will be selected for this study (randomized and double blind) and divided into 3 groups (n = 25): Group 1 - Pulse Laser (880nm, 30mW, 3,6J / cm², 25Hz) ; Group 2 - Continuous Laser (880nm; 30mW; 3.6J / cm²); Group 3 - Placebo. The efficacy of the laser will be assessed using the VAS scale 10 minutes after the laser application, immediately before the blockade is performed.

DETAILED DESCRIPTION:
Anxiety, pain and discomfort are situations of great stress in the daily routine of clinical practice, and especially in the practice of the dental emergency sector. Several studies have concluded that low-intensity laser therapy has been shown to be effective in pain management. However, the majority report the use of laser in the treatment of chronic pain, few studies show its application in acute pain and only one study evaluated the effect of low laser on acute pain of pulp inflammation, but with other parameters. In addition, because of the inflammatory process and several factors of unknown origin, the anesthetic agent can not always promote complete analgesia, especially when faced with mandibular molars. Therefore, the present study has the objective of evaluating whether the previous therapy with low intensity laser, through its analgesic effect, can promote a greater comfort specifically for this type of patient. 75 patients with pain from mandibular molar pulpitis will be selected for this study (randomized and double blind) and divided into 3 groups (n = 25): Group 1 - Pulse Laser (880nm, 30mW, 3,6J / cm², 25Hz) ; Group 2 - Continuous Laser (880nm; 30mW; 3.6J / cm²); Group 3 - Placebo. The pain will be evaluated by means of an VAS score in 6 different times: initial pain, immediately after and 10 minutes after irradiation with the laser, 10 minutes after inferior alveolar nerve block (IANB), during conventional endodontic treatment, after the end of the procedure. (T0, T1, T1 ', T2, T3 and T4). The efficacy of the laser application will be assessed using the VAS scale 10 minutes after the laser application, immediately before the blockade is performed. The use of the laser will be considered effective if the patient reports a reduction in the VAS scale of 2 points, between the initial moment and 10 minutes after the laser application. Analgesia will be evaluated during the pulpectomy procedure with the use of the verbal analogue scale 0 to 3. Analgesic effect will be considered if the professional can finish the procedure without the patient reporting 2 or 3 on this scale. The data obtained between the different groups and schedules will be compared statistically, and the statistical test chosen will depend on the normality of the data. The data obtained between the different groups and times will be compared statistically, and the statistical test chosen will depend on the normality of the data.

ELIGIBILITY:
Inclusion Criteria:

* ASA I patients, according to the classification of the American Society of Anesthesiology (ASA)
* 18 and 50 years
* Systolic pressure below 140 mmHg and diastolic below 90 mmHg and heart rate between 70 - / + 20 beats / minute
* Pulpectomy in the first and / or lower second molars, which has at least one adjacent molar tooth and a contralateral canine; or absence of deep cavities, extensive restorations, advanced periodontal disease and no history of trauma or sensitivity.

Exclusion Criteria:

* Patients with a history of sensitivity to local anesthetics and sulfur
* Pregnant or suspected of pregnancy
* Users of medications that may interact with the local anesthetic, such as, anxiolytics, antidepressants, antipsychotics, β-blockers and antihistaminic agents
* Patients with septic process near the injection site
* Patients under orthodontic treatment
* Patients with heart disease, neurological disease, hyperthyroidism and diabetes; drug users.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction in VAS score | 10 minutes
  The success of laser use was defined as a reduction of more than 2 in the patient's pain report between the initial moment and 10 minutes after the laser application

SECONDARY OUTCOMES:
Analgesia | 30 minutes
  The success of IANB associated with laser therapy will be defined as the ability to access the pulp chamber and perform the pulpectomy without the pain being classified as uncomfortable by the patient (0 to 1 scale) during the treatment,which takes almost 30 minutes to be completed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramalho KM, de Souza LM, Tortamano IP, Adde CA, Rocha RG, de Paula Eduardo C. A randomized placebo-blind study of the effect of low power laser on pain caused by irreversible pulpitis. Lasers Med Sci. 2016 Dec;31(9):1899-1905. doi: 10.1007/s10103-016-2068-7. Epub 2016 Oct 1. PMID 27696017